CLINICAL TRIAL: NCT05005104
Title: Predictors of Complicated Appendicitis Among Patients Presented to Public Referral Hospitals in Harari Region: A Case-control Study
Brief Title: Causes of Complicated Appendicitis at Referral Hospital
Acronym: AA
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Badhaasaa, Dr, Haramaya Unversity
Other Study IDs: IHRERC/005/2021
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Complicated Appendicitis
Keywords: complicated appendicitis, acute abdomen
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was conducted on a medical record of previously treated patients for acute appendicitis at HFSUH, Harar, Ethiopia. The study design was case-control with a total sample size of 402.

DETAILED DESCRIPTION:
The case-control study conducted at HFSUH was proceeded following the university's protocol and after passing institutional ethical review permission.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with acute appendicitis

Exclusion Criteria:

* incidental appendectomy patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with a diagnosis of acute appendicitis and admitted to a public hospital in Harari regional state.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Number of patients having the predictors of complicated appendicitis. | 1 week
  Clinical histories like duration of chief complaint, constipation, vomiting, fever, visiting to lower level clinics, presence of comorbidities were used to assess the factors associated with complicated appendicitis.

CONTACTS AND LOCATIONS:
Overall Officials: Badhaasaa Bayissa, MD, Principal Investigator — HU
Locations (1):
- CHMS, Harar, Harari NS, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
on reasonable request